CLINICAL TRIAL: NCT04921891
Title: Comparison of Block Success in Patients Undergoing Ultrasound-guided Infraclavicular Brachial Plexus Block With Bilateral Upper Extremity Perfusion Index
Brief Title: Is Perfusion Index an Indicator of Block Success in Ultrasound-guided Infraclavicular Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Gokhan Sertcakacilar, MD, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2014-86
Record Dates: First submitted 2021-06-01; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Carpal Tunnel Syndrome; Perfusion Index
Keywords: Infraclavicular block; Perfusion index; Ultrasonography; Block assessment
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Nerve Block

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blocked arm (Active Comparator): The investigators performed an infraclavicular nerve block to the operated arm group to provide anesthesia.
  Interventions: Procedure: Infraclavicular nerve block
- Unblocked arm (Active Comparator): The upper extremity without block was assigned as the control group, and a comparison was made between the two upper extremities.
  Interventions: Procedure: Without nerve block

INTERVENTIONS:
Procedure: Infraclavicular nerve block — The investigators performed an infraclavicular nerve block to the operated arm group to provide anesthesia.
  Arms: Blocked arm
Procedure: Without nerve block — The upper extremity without block was assigned as the control group, and a comparison was made between the two upper extremities.
  Arms: Unblocked arm

SUMMARY:
The infraclavicular nerve block, which is frequently preferred in upper extremity surgeries, provides additional advantages such as reduction in opioid consumption by providing analgesic effect in the postoperative period as welll. The success of peripheral nerve blocks is usually assessed by subjective feedback from the patient, and patient cooperation is needed. The aim of this study is to assess whether the perfusion index level, which can be measured noninvasively, can be a predictor of the infraclavicular block success.

DETAILED DESCRIPTION:
Thirty patients who were operated on for carpal tunnel syndrome under infraclavicular brachial plexus block were included in our study. After the procedure, at 10-minute intervals, the sensory block was assessed by a pinprick test, and the motor block was assessed by the ability to flex the hand and the forearm. In addition, PI and skin temperature were measured 0-10-20-30 minutes after the block and at postoperative 2, 4, and 6 hours. 30 minutes after the measurements, the surgical procedure was allowed to begin in patients with successful block.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18-75
* Patients who will diagnose with carpal tunnel syndrome by electroneuromyography (ENMG), and will undergo unilateral surgery under elective conditions
* ASA I-II-III patients

Exclusion Criteria:

* Patients who will refuse this method
* Neurological deficits,
* Diabetes mellitus,
* Local anesthetic allergy,
* Morbidly obese,
* Peripheral vascular disease, coronary artery disease, or coagulopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04-15 (Actual); Primary Completion 2014-04-15 (Actual); Study Completion 2014-10-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of whether perfusion index is a reliable and objective method to indicate block success | 6 hours postprocedurly
  Perfusion index was measured up to 6 hours after the procedure.

SECONDARY OUTCOMES:
Determining of a cut-off value for PI and PI ratio for a successful block. | Up to 6 hours after the procedure
  There may be changes in the cut-off value depending on the applied plexus area, local anesthesia, volume and concentration of LA and the applied assistive technique (ultrasound or nerve stimulator). For both this reason and due to the high variability in the PI values, the PI ratio was calculated to predict block success.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Bakirkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided